CLINICAL TRIAL: NCT03131167
Title: A Randomized, Double-masked, Placebo-controlled Phase 1 Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single Daily and Multiple Daily Ascending Doses of SHP639 Topical Ophthalmic Solution in Subjects With Ocular Hypertension or Primary Open-angle Glaucoma (POAG)
Brief Title: Study of SHP639 Eye Drops in Adults With High Eye Pressure or Primary Open-angle Glaucoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHP639-101
Record Dates: First submitted 2017-04-20; First posted 2017-04-27 (Actual); Results first posted 2019-08-07 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-05

CONDITIONS: Primary Open-angle Glaucoma (POAG); Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SHP639 Ophthalmic Solution Arm (n=60) (Experimental): Participants are divided into groups called cohorts. There will be approximately 12 cohorts, each consisting of 7 participants. In each cohort 5 out of 7 participants will be assigned a specified concentration of SHP639 (0.1%, 0.3%, or 0.6%) ophthalmic solution and a specific dosing schedule (the study participants will be instructed to insill the study drug one, two, three, or four times a day) in both eyes during the study.
  Interventions: Drug: SHP639 (n=60)
- Vehicle Ophthalmic Arm (n=24) (Placebo Comparator): In each cohort 2 out of 7 participants will be assigned a placebo ophthalmic solution matched to 0.1%, 0.3%, and 0.6% SHP639 ophthalmic solution and specific dosing schedule (the study participants will be instructed to instill the study drug one, two, three, or four times a day) in both eyes during the study.
  Interventions: Drug: Placebo Comparator (n=24)

INTERVENTIONS:
Drug: SHP639 (n=60) — Drug SHP639 is a 9-amino acid, synthetic, C-type natriuretic peptide (CNP) analog.
  Arms: SHP639 Ophthalmic Solution Arm (n=60)
Drug: Placebo Comparator (n=24) — Drug: Vehicle Ophthalmic placebo solution of the same composition as the test product.
  Arms: Vehicle Ophthalmic Arm (n=24)

SUMMARY:
Safety and tolerability of three different concentrations (0.1%, 03%, 0.6%) of the investigational SHP639 eye drops will be evaluated in participants with high eye pressure or primary open-angle glaucoma.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must provide written, signed and dated informed consent to participate in the study in accordance with the International Council for Harmonisation (ICH) Good Clinical Practice (GCP) Guideline E6(R1) and applicable regulations, before completing any study-related procedures.
2. Participants must be aged from 18 through 90 at the time of consent. This inclusion criterion will only be assessed at the screening visit.
3. Participants must have ocular hypertension (OHT) or stable early primary open-angle glaucoma (POAG) in both eyes with acceptable Humphrey visual fields (HVF). Early POAG for this protocol is defined as healthy appearing anterior chamber angles (Shaffer classification system grade 3 or 4) and focal and/or generalized thinning of the optic disc rim characteristic of glaucomatous disease. An acceptable HVF must have been performed within approximately one year of screening, have a false-positive rate of 25 percent (%) maximum, false-negative rate of 25% maximum, and fixation loss rate of 33% maximum, and mean deviation of no worse than -6.00 decibels (dB).
4. On Day -1, participants must have a mean IOP of greater than or equal to (>=) 24 millimeter of mercury (mmHg) at 8:00 AM and a mean IOP of >= 22 mmHg at 10:00 AM in at least 1 eye, with an IOP difference of less than (<) 4 mmHg between eyes at both of these time points. If only 1 eye meets this criterion, then it will be the designated study eye for pharmacodynamic analysis; this eye will also be used for dosing in Cohort A single-dose treatment period (SDTP).
5. Participants must have a best-corrected visual acuity (BCVA) in both eyes of 65 letters on the Early Treatment Diabetic Retinopathy Study chart (Snellen equivalent approximately [∼] 20/60) or better at the screening and baseline assessments.
6. Participants must be males or females who are non-pregnant and non-lactating at screening (negative serum beta-human chorionic gonadotropin [beta-hCG]); if sexually active during the study, they must agree to comply with the applicable contraceptive requirements throughout the study period and for 60 days following the last dose of investigational product.
7. Participants must have a satisfactory medical assessment with no clinically significant or relevant abnormalities as determined by medical history, physical examination, and clinical and laboratory evaluation (hematology, biochemistry, urinalysis) as assessed by the investigator.
8. Participants must understand and be able, willing, and likely to fully comply with study procedures and restrictions.
9. Participants must be non-smokers or have had stable use of tobacco or nicotine-containing products for a 3-month period before signing the informed consent form (ICF).
10. Participants who drink alcohol must have had stable use of alcohol for a 3-month period before signing the ICF.

Exclusion Criteria:

1. Participant has an anatomically narrow angle, synechiae or evidence of prior inflammation, angle closure glaucoma, normal tension glaucoma, pseudoexfoliation syndrome or pigmentary dispersion syndrome with or without glaucoma, or secondary glaucoma.
2. Participant has corneal endothelial cell counts of less than 2000 cells per millimeter^2 (measured by noncontact specular microscopy) at the screening or baseline assessments.
3. Participant has central corneal thickness less than 500 micrometer (mcm) or greater than 620 mcm at the screening or baseline assessments.
4. Participant has IOP greater than 32 mmHg in either eye before randomization.
5. Participant has used topical ocular hypotensive medications as follows: prostaglandin analogs, beta-adrenoceptor antagonists, alpha-adrenergic agonists, or epinephrine-related medications within 4 weeks before the first dose of investigational product; or pilocarpine or carbonic anhydrase inhibitors within 7 days before the first dose of investigational product.
6. Participant has a history of angle closure, ocular surgery, microinvasive glaucoma surgery device insertion, or laser surgery, except for the following procedures, which are allowed: uncomplicated cataract surgery, laser peripheral iridotomy with resultant angle of Shaffer grade 3 or 4, and postcataract neodymium-doped yttrium-aluminum-garnet (Nd:YAG) laser posterior capsulotomy. Cataract surgery and other procedures must have occurred a minimum of 3 months before randomization.
7. Participant has a history of significant ocular trauma or ocular disease including but not limited to moderate to severe dry eye disease that requires chronic treatment or punctal plugs.
8. Participant has evidence of ocular infection, inflammation, degeneration, or dystrophy at the screening or baseline assessments, including but not limited to moderate to severe blepharitis (mild blepharitis is allowed), conjunctivitis (allergic or infectious), corneal dystrophy (epithelial, stromal, or endothelial), corneal haze of grade 1 or greater based on the Hwang Grading Scale of Corneal Haze, corneal opacities, keratitis, uveitis, or vitritis.
9. Participant has retinal disease including but not limited to: moderate or severe non-proliferative diabetic retinopathy (NPDR) (early NPDR is allowed), proliferative diabetic retinopathy, intermediate or advanced dry age-related macular degeneration (AMD) (early dry AMD is allowed), all geographic atrophy, or all wet AMD.
10. Participant has any non-glaucomatous optic neuropathy or other significant non-glaucomatous ocular disease that is likely to affect visual function.
11. Participant has any corneal or ocular surface pathology in either eye that prevents proper IOP measurement, pachymetry, or other study data collection procedures.
12. Participant has had changes to their existing prescription medication regimen for chronic disease, including those medicines that affect IOP, within 14 days or 5 half-lives before screening, whichever is longer.
13. Participant has started any new prescription drug medication for chronic disease, including those medicines that affect IOP, within 14 days or 5 half-lives before screening, whichever is longer.
14. Participant has a history of corticosteroid use within 3 months before randomization, except for non-periocular dermatologic use, which is allowed.
15. Participant has used belladonna alkaloids (scopolamine, hyoscamine, atropine) within 7 days prior to randomization, cannabinoids or opioids within 28 days before randomization, or B-type natriuretic peptides within the past year before randomization; or a participant has an anticipated need for any of the aforementioned drugs/drug categories during the study.
16. Participant has used amantadine within 28 days before randomization.
17. Participant is unable to discontinue contact lens use during and for 60 minutes following instillation of study medication, during ophthalmologic examinations, and during study visits.
18. Participant has a current or relevant history of any physical, medical, mental, or psychiatric illness, disorder, or condition that may require treatment during the study and/or that may interfere with the participant complying with the study rules and procedures or completing the study.
19. Participant has any condition that presents undue risk from use of the investigational product, assessment tools, or procedures.
20. Participant is a woman who is pregnant (positive serum beta-hCG pregnancy test at the time of screening), lactating, or less than 90 days post-partum at randomization.
21. Participant has donated blood within 60 days before first dose of investigational product.
22. Participant has donated plasma within 28 days before first dose of investigational product.
23. Participant has used another investigational product within 30 days before the first dose of investigational product or is actively enrolled in a drug or vaccine clinical study.
24. Participant has a positive human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV) antibodies screen.
25. Participant has a positive drugs of abuse screen or alcohol breathalyzer test.
26. Participant has been previously enrolled in this study.
27. Participant has known hypersensitivity or allergy to any of the ingredients of the investigational product.
28. Participant consumes more than 21 units of alcohol per week or is unable to refrain from alcohol consumption within 48 hours before a scheduled visit. (1 alcohol unit=1 beer or 1 wine [5 ounce per 150 milliliter] or 1 liquor [1.5 ounce per 40 milliliter] or 0.75 ounce alcohol.)
29. Participant is unable to refrain from tobacco or any products containing nicotine within 8 hours before a scheduled visit.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2017-05-10 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Central Contact, Lexington, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 4 study centers in the United States between 10 May 2017 (first participant first visit) and 30 May 2018 (last participant last visit).
Pre-assignment Details: Totally, 63 participants enrolled, randomized and received treatment in two parts of the study with one cohort for one dose level (Part 1: Cohort A1, A2, A3, with single dose and QD multiple dose, followed by Cohort B1, B2, B3 with BID multiple dose. Part 2: Cohort C1, C2, C3 with TID multiple dose, followed by D1, D2, D3 with QID multiple dose).
Groups:
- Placebo QD: Participants received one drop of placebo matched to SHP639 at a dose of 0.1%, 0.3%, 0.6% respectively applied topically in the designated eye once daily (QD) during the once daily dose regimen.
- SHP639 0.1% QD: Participants received one drop of SHP639 at a dose of 0.1% applied topically in the designated eye once daily (QD) during the once daily dose regimen.
- SHP639 0.3% QD: Participants received one drop of SHP639 at a dose of 0.3% applied topically in the designated eye once daily (QD) during the once daily dose regimen.
- SHP639 0.6% QD: Participants received one drop of SHP639 at a dose of 0.6% applied topically in the designated eye once daily (QD) during the once daily dose regimen.
- Placebo BID: Participants received one drop of placebo matched to SHP639 at a dose of 0.1%, 0.3%, 0.6% respectively applied topically in the designated eye and non study eye twice daily (BID) during the twice daily dose regimen.
- SHP639 0.1% BID: Participants received one drop of SHP639 at a dose of 0.1% applied topically in the designated eye and non study eye twice daily (BID) during the twice daily dose regimen.
- SHP639 0.3% BID: Participants received one drop of SHP639 at a dose of 0.3% applied topically in the designated eye and non study eye twice daily (BID) during the twice daily dose regimen.
- SHP639 0.6% BID: Participants received one drop of SHP639 at a dose of 0.6% applied topically in the designated eye and non study eye twice daily (BID) during the twice daily dose regimen.
- Placebo Repeated BID: Participants received one drop of placebo matched to SHP639 at a dose of 0.6% applied topically in the designated eye and non study eye twice daily (BID) during the repeated twice daily dose regimen.
- SHP639 0.6% Repeated BID: Participants received one drop of SHP639 at a dose of 0.6% applied topically in both the designated eye and non study eye twice daily (BID) during the repeated twice daily dose regimen.
- Placebo TID: Participants received one drop of placebo matched to SHP639 at a dose of 0.1%, 0.3%, 0.6% respectively applied topically in the designated eye and non study eye thrice daily (TID) during the thrice daily dose regimen.
- SHP639 0.1% TID: Participants received one drop of SHP639 at a dose of 0.1% applied topically in the designated eye and non study eye thrice daily (TID) during the thrice daily dose regimen.
- SHP639 0.3% TID: Participants received one drop of SHP639 at a dose of 0.3% applied topically in the designated eye and non study eye thrice daily (TID) during the thrice daily dose regimen.
Period: Overall Study
Arm/Group | Placebo QD | SHP639 0.1% QD | SHP639 0.3% QD | SHP639 0.6% QD | Placebo BID | SHP639 0.1% BID | SHP639 0.3% BID | SHP639 0.6% BID | Placebo Repeated BID | SHP639 0.6% Repeated BID | Placebo TID | SHP639 0.1% TID | SHP639 0.3% TID
Started | 6 | 5 | 5 | 5 | 6 | 5 | 5 | 5 | 2 | 5 | 4 | 5 | 5
Completed | 6 | 5 | 5 | 5 | 6 | 4 | 5 | 5 | 2 | 5 | 4 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other (Unspecified) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Randomized set consisted of all participants in the enrolled set for whom a randomization number was assigned.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo QD | SHP639 0.1% QD | SHP639 0.3% QD | SHP639 0.6% QD | Placebo BID | SHP639 0.1% BID | SHP639 0.3% BID | SHP639 0.6% BID | Placebo Repeated BID | SHP639 0.6% Repeated BID | Placebo TID | SHP639 0.1% TID | SHP639 0.3% TID | Total
Number analyzed (Participants) | 6 | 5 | 5 | 5 | 6 | 5 | 5 | 5 | 2 | 5 | 4 | 5 | 5 | 63
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.0 (7.77) | 63.8 (7.46) | 67.6 (6.39) | 59.0 (2.74) | 68.7 (8.19) | 72.8 (8.58) | 69.0 (7.31) | 68.2 (6.69) | 70.0 (4.24) | 74.6 (5.18) | 67.5 (18.38) | 70.8 (14.04) | 69.4 (4.93) | 68.4 (8.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 2 | 4 | 5 | 5 | 2 | 4 | 0 | 4 | 2 | 3 | 4 | 43
  Male | 2 | 1 | 3 | 1 | 1 | 0 | 3 | 1 | 2 | 1 | 2 | 2 | 1 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 4 | 7
  Not Hispanic or Latino | 6 | 5 | 5 | 5 | 5 | 5 | 4 | 5 | 2 | 5 | 3 | 5 | 1 | 56
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 5 | 1 | 5 | 2 | 0 | 5 | 2 | 0 | 0 | 0 | 0 | 0 | 24
  White | 2 | 0 | 3 | 0 | 4 | 4 | 0 | 3 | 2 | 5 | 4 | 5 | 5 | 37
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Event (TEAE)
Description: An adverse event (AE) is any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. TEAEs were defined as AEs with a start date on or after the first dose of double-blind investigational product or a start date before the date of the first dose of double-blind investigational product that increased in severity or after the date of the first dose.
Time Frame: From start of study drug administration up to follow-up (Day 88)
Population: Safety set consisted of all participants who were randomized and who received at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo QD | SHP639 0.1% QD | SHP639 0.3% QD | SHP639 0.6% QD | Placebo BID | SHP639 0.1% BID | SHP639 0.3% BID | SHP639 0.6% BID | Placebo Repeated BID | SHP639 0.6% Repeated BID | Placebo TID | SHP639 0.1% TID | SHP639 0.3% TID
Number analyzed (Participants) | 6 | 5 | 5 | 5 | 6 | 5 | 5 | 5 | 2 | 5 | 4 | 5 | 5
Participants | 2 | 0 | 2 | 0 | 2 | 2 | 0 | 5 | 1 | 5 | 2 | 1 | 3

2. Secondary Outcome: Change From Baseline in Intra Ocular Pressure (IOP) at Day 29
Description: IOP was measured using Goldmann applanation tonometry and reported data from baseline at day 29 for both study eye and non study eye.
Time Frame: Baseline, Day 29
Population: Pharmacodynamic (PD) set consisted of all participants in the safety set for whom the primary PD data were evaluable.
Measure: Mean (Standard Deviation); unit: millimeter of mercury (mmHg)
Arm/Group | Placebo QD | SHP639 0.1% QD | SHP639 0.3% QD | SHP639 0.6% QD | Placebo BID | SHP639 0.1% BID | SHP639 0.3% BID | SHP639 0.6% BID | Placebo Repeated BID | SHP639 0.6% Repeated BID | Placebo TID | SHP639 0.1% TID | SHP639 0.3% TID
Number analyzed (Participants) | 6 | 5 | 5 | 5 | 6 | 5 | 5 | 5 | 2 | 5 | 4 | 5 | 5
millimeter of mercury (mmHg)
  Study Eye | 0.00 (1.294) | -1.20 (1.605) | 0.45 (1.515) | 0.40 (1.084) | 0.38 (1.539) | 0.44 (1.972) | -0.20 (0.837) | -0.40 (2.826) | -0.13 (2.652) | -2.00 (1.490) | -1.13 (4.539) | 0.10 (0.929) | -4.65 (3.170)
  Non-Study Eye | -0.38 (1.430) | -1.50 (0.354) | 1.20 (2.087) | 0.70 (0.908) | 0.83 (1.393) | 0.50 (1.061) | -0.20 (0.758) | -0.25 (2.610) | -1.00 (4.243) | -1.80 (2.260) | 0.00 (3.889) | -0.10 (1.421) | -3.85 (2.389)

ADVERSE EVENTS:
Time Frame: From start of study drug administration up to follow-up (day 88)
Arm/Group | Placebo QD | SHP639 0.1% QD | SHP639 0.3% QD | SHP639 0.6% QD | Placebo BID | SHP639 0.1% BID | SHP639 0.3% BID | SHP639 0.6% BID | Placebo Repeated BID | SHP639 0.6% Repeated BID | Placebo TID | SHP639 0.1% TID | SHP639 0.3% TID
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/5 | 0/5 | 0/5 | 0/6 | 0/5 | 0/5 | 0/5 | 0/2 | 0/5 | 0/4 | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/5 | 0/5 | 0/5 | 0/6 | 0/5 | 0/5 | 0/5 | 0/2 | 0/5 | 0/4 | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 2/6 | 0/5 | 2/5 | 0/5 | 2/6 | 2/5 | 0/5 | 5/5 | 1/2 | 5/5 | 2/4 | 1/5 | 3/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo QD (N=6) | SHP639 0.1% QD (N=5) | SHP639 0.3% QD (N=5) | SHP639 0.6% QD (N=5) | Placebo BID (N=6) | SHP639 0.1% BID (N=5) | SHP639 0.3% BID (N=5) | SHP639 0.6% BID (N=5) | Placebo Repeated BID (N=2) | SHP639 0.6% Repeated BID (N=5) | Placebo TID (N=4) | SHP639 0.1% TID (N=5) | SHP639 0.3% TID (N=5)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abnormal sensation in eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctival hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Eye discharge (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye disorder (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye pruritus (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eyelid margin crusting (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Instillation site discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Instillation site pain (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (7) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vital dye staining cornea present (Investigations) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 5 (7) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.

DOCUMENTS (2):
  • Study Protocol (2018-05-11): https://cdn.clinicaltrials.gov/large-docs/67/NCT03131167/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-30): https://cdn.clinicaltrials.gov/large-docs/67/NCT03131167/SAP_001.pdf